CLINICAL TRIAL: NCT05111028
Title: Reversal of Aspirin Antiplatelet Therapy With Cold Stored Platelets
Acronym: RASP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bloodworks (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Reversal of Platelet Aggregation Inhibitors
Keywords: Aspirin; Blood Platelets; Platelet Aggregation Inhibitors; Platelet Transfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Active Comparator): Each research subject will participate in two study periods that will crossover from one storage product to the other storage product (Cold Stored Platelets vs Room Temperature Platelets) based on the randomization assignment. In Period 1 subjects will undergo an apheresis platelet collection, aspirin dosing, transfusion of their autologous platelets, and followed by platelet response testing and safety assessments. This is repeated in Period 2 using the other storage product. CSP is the the experimental comparator and RTP is the active comparator.
  Interventions: Biological: Autologous Room Temperature stored Platelet transfusion; Biological: Autologous Cold Stored Platelet transfusion
- Period 2 (Experimental): Each research subject will participate in two study periods that will crossover from one storage product to the other storage product (Cold Stored Platelets vs Room Temperature Platelets) based on the randomization assignment. In Period 1 subjects will undergo an apheresis platelet collection, aspirin dosing, transfusion of their autologous platelets, and followed by platelet response testing and safety assessments. This is repeated in Period 2 using the other storage product. CSP is the the experimental comparator and RTP is the active comparator.
  Interventions: Biological: Autologous Room Temperature stored Platelet transfusion; Biological: Autologous Cold Stored Platelet transfusion

INTERVENTIONS:
Biological: Autologous Room Temperature stored Platelet transfusion — An autologous transfusion of platelets stored at 22°C for 7 days.
Biological: Autologous Cold Stored Platelet transfusion — An autologous transfusion of platelets stored at 4°C for 7, 14, 21, or 28 days.

SUMMARY:
Purpose of this study is to compare the reversal responses of 4°C cold stored platelets (CSP) versus 7 day, 22°C room temperature stored platelets (RTP) when given to healthy adult subjects who have received a loading dose of aspirin antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject feels healthy and well
* 18-59 years old
* All sexes
* Temperature <99.6 F
* Resting blood pressure: systolic <181 mmHg, diastolic <101 mmHg
* Resting heart rate: 40 - 100 beats per minute
* Weight: >109 lb
* Hematocrit: >34% for female subjects, >37% for male subjects. <56% for all subjects.
* Platelet count able to achieve target platelet yield per apheresis machine configuration parameters
* Subjects must be able to read, understand and sign the informed consent document and commit to the study follow-up schedule. The ability to read and speak English is required for participation
* Subject must agree to avoid taking any aspirin or aspirin-containing drugs (e.g., Alka-Seltzer®, Bufferin®, Excedrin®) or NSAIDs (e.g.,Feldene®, Motrin®, Aleve®, Advil®) or other drugs known to significantly affect platelet function throughout their study participation determined by PI
* Subjects must have "good veins" for apheresis platelet collection and drawing blood samples
* Women of child-bearing potential must agree to use an effective method of contraception during the course of the study. The following methods of contraception will be considered 'effective' when self-reported by subject; abstinence, intrauterine contraception devices, hormonal methods, barrier methods or history of sterilization
* Subject has phone and e-mail for contact and notification, and is able to come to the research site for study visits

Exclusion Criteria:

1. Active acute infection or suspected active infection or taking antibiotics.
2. Active immune/inflammatory condition (e.g. gout, systemic lupus erythematosus, allograft rejection).
3. History of heart disease, including endorsement of shortness of breath with mild exertion (at the discretion of the PI).
4. History of significant liver, kidney, GI, blood, endocrine/metabolic, autoimmune or pulmonary disease, untreated hypertension and or metabolic syndrome (at the discretion of the PI).
5. Diabetes Mellitus.
6. Cancer of any kind (exceptions being basal or squamous cell cancers of the skin), under treatment or resolved.
7. History of bleeding events, family history of bleeding events, or known genetic disorder with bleeding diathesis.
8. A family history of venous or arterial thrombosis before the age of 50 in first degree relatives.
9. A personal history of DVT, venous or arterial thrombosis, blood clots or stroke.
10. History of or currently prescribed antiplatelet therapies [such as clopidogrel (Plavix), ticlopidine (Ticlid) or Ticagrelor (Brilinta)] and/or anticoagulant therapies [such as heparin, enoxaparin (Lovenox), warfarin (Coumadin), apixaban (Eliquis), dabigatran (Pradaxa), edoxaban (Savaysa), rivaroxaban (Xarelto)].
11. Subject has taken any aspirin or aspirin-containing drugs (e.g., Alka-Seltzer®, Bufferin®, Excedrin®) or NSAIDs (e.g.,Feldene®, Motrin®, Aleve®, Advil®) or other drugs known to significantly affect platelet function within 14 days prior to screening as determined by PI.
12. Chronic NSAID therapy.
13. Chronic steroid therapy.
14. Known allergy to aspirin.
15. Current drug or alcohol dependence by subject's declaration.
16. Currently pregnant or nursing as assessed during interview. A urine pregnancy test prior to apheresis is required for women of childbearing potential.
17. Subject plans to participate in contact sports during study/observational period such as boxing, rugby, American football, soccer, or other risky recreational hobbies at the discretion of the investigator.
18. Unwilling or unable to comply with the protocol in the opinion of the investigator.
19. Participation in an experimental drug/device study within the past 30 days (other than this study). Subjects who have received an infusion on this study may not be re-enrolled.
20. Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Glycoprotein IIb/IIIa activation at 1hr post transfusion | 1 hour after autologous transfusion
  The primary endpoint is αIIbβ3 (GPIIb-IIIa) integrin activation determined by ARU (Verify Now Aspirin [ARUTest]) at 1h post autologous transfusion

SECONDARY OUTCOMES:
Glycoprotein IIb/IIIa activation at 4hr post transfusion | 4 hours after autologous transfusion
  A secondary endpoint is αIIbβ3 (GPIIb-IIIa) integrin activation determined by ARU (Verify Now Aspirin [ARUTest]) at 4h post autologous transfusion
Glycoprotein IIb/IIIa activation at 24hr post transfusion | 24 hours after autologous transfusion
  A secondary endpoint is αIIbβ3 (GPIIb-IIIa) integrin activation determined by ARU (Verify Now Aspirin [ARUTest]) at 24h post autologous transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Stolla, MD, PhD, Principal Investigator — Bloodworks
Locations (1):
- Bloodworks Northwest Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Your data or specimens collected as part of this research will not be used for future research studies or given to anyone else for future research studies, even if all information that personally identifies you is removed.